CLINICAL TRIAL: NCT06493760
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of SSGJ-707 As First-Line Treatment in Metastatic Colorectal Cancer Patients
Brief Title: A Phase 2 Study of SSGJ-707 in Metastatic Colorectal Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-707-CRC-II-01
Record Dates: First submitted 2024-06-25; First posted 2024-07-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: SSGJ-707; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- SSGJ-707(dose 1)+ XELOX (Experimental)
  Interventions: Drug: SSGJ-707; Drug: Oxaliplatin; Drug: Capecitabine
- SSGJ-707(dose 1)+ mFOLFOX6 (Experimental)
  Interventions: Drug: SSGJ-707; Drug: Oxaliplatin; Drug: Calcium Folinate; Drug: 5-fluorouracil
- SSGJ-707(dose 2)+ XELOX (Experimental)
  Interventions: Drug: SSGJ-707; Drug: Oxaliplatin; Drug: Capecitabine
- SSGJ-707(dose 2)+ mFOLFOX6 (Experimental)
  Interventions: Drug: SSGJ-707; Drug: Oxaliplatin; Drug: Calcium Folinate; Drug: 5-fluorouracil
- SSGJ-707+XELOX/mFOLFOX6 (Experimental)
  Interventions: Drug: SSGJ-707; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Calcium Folinate; Drug: 5-fluorouracil
- Bevacizumab+XELOX/mFOLFOX6 (Active Comparator)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Calcium Folinate; Drug: 5-fluorouracil
- SSGJ-707 monotherapy (Experimental)
  Interventions: Drug: SSGJ-707

INTERVENTIONS:
Drug: SSGJ-707 — bispecific antibody
  Arms: SSGJ-707 monotherapy; SSGJ-707(dose 1)+ XELOX; SSGJ-707(dose 1)+ mFOLFOX6; SSGJ-707(dose 2)+ XELOX; SSGJ-707(dose 2)+ mFOLFOX6; SSGJ-707+XELOX/mFOLFOX6
Drug: Bevacizumab — VEGF antibody
  Arms: Bevacizumab+XELOX/mFOLFOX6
Drug: Oxaliplatin — chemotherapy
  Arms: Bevacizumab+XELOX/mFOLFOX6; SSGJ-707(dose 1)+ XELOX; SSGJ-707(dose 1)+ mFOLFOX6; SSGJ-707(dose 2)+ XELOX; SSGJ-707(dose 2)+ mFOLFOX6; SSGJ-707+XELOX/mFOLFOX6
Drug: Capecitabine — chemotherapy
  Arms: Bevacizumab+XELOX/mFOLFOX6; SSGJ-707(dose 1)+ XELOX; SSGJ-707(dose 2)+ XELOX; SSGJ-707+XELOX/mFOLFOX6
Drug: Calcium Folinate — chemotherapy
  Arms: Bevacizumab+XELOX/mFOLFOX6; SSGJ-707(dose 1)+ mFOLFOX6; SSGJ-707(dose 2)+ mFOLFOX6; SSGJ-707+XELOX/mFOLFOX6
Drug: 5-fluorouracil — chemotherapy
  Arms: Bevacizumab+XELOX/mFOLFOX6; SSGJ-707(dose 1)+ mFOLFOX6; SSGJ-707(dose 2)+ mFOLFOX6; SSGJ-707+XELOX/mFOLFOX6

SUMMARY:
This study includes two parts:Part 1: SSGJ-707 (different dosing regimens) in combination with chemotherapy for first-line treatment of metastatic colorectal cancer.Part 2: SSGJ-707 in combination with chemotherapy versus bevacizumab in combination with chemotherapy for first-line treatment of metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented metastatic colorectal cancer confirmed .
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >=12 weeks.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to SSGJ-707 The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 months
  Objective response rate
Safety and tolerability | 12 months
  Safety and tolerability assessed by incidence and severity of adverse events

SECONDARY OUTCOMES:
PFS | 24 months
  The efficacy end points

CONTACTS AND LOCATIONS:
Locations (1):
- Liu Tianshu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No